CLINICAL TRIAL: NCT03661294
Title: Feasibility Study to Investigate the Energy Expenditure of Acute Spinal Cord Injured Patients at Different Stages of Rehabilitation
Brief Title: Investigating the Energy Expenditure of Acute Spinal Cord Injured Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Nutricia UK Ltd (Industry); University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STH18054
Record Dates: First submitted 2017-07-13; First posted 2018-09-07 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Spinal Cord Injury, Acute
Keywords: Energy, spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GE Healthcare Metabolic Oxygenator (Other): The actual and predicted energy expenditure of tetraplegic (ventilated/non-vent) and paraplegic patients will be measured at three time points during the patient's rehabilitation in hospital.
  Interventions: Diagnostic Test: GE Healthcare Metabolic Oxygenator

INTERVENTIONS:
Diagnostic Test: GE Healthcare Metabolic Oxygenator

SUMMARY:
It is recognised that weight gain is a common problem in patients with a spinal cord injury and can lead to an increased incidence of metabolic syndrome. Weight gain is thought to be attributed to excess calorie intake, reduction in energy requirements and / or a reduction in exercise. However, further understanding of this energy imbalance needs to be addressed.

This feasibility study will initially determine if it is feasible to measure the 'actual' energy requirements of 15 paraplegic and 15 tetraplegic (ventilated and non-ventilated) in-patients during bed rest and rehabilitation following acute SCI. This preliminary data will be compared to 'predicted' energy expenditure levels. The calorie intake and body composition for each patient will be measured as well as factors indicative of metabolic syndrome. The study will initially provide statistical information in order to estimate the sample size required for a future definitive study.

DETAILED DESCRIPTION:
Introduction:

There are an estimated 40,000 people living with a Spinal Cord Injury (SCI) in the UK alone (http://www.apparelyzed.com/statistics.html). Although there have been improvements in medical care, mortality rates are still elevated compared to the able-bodied population. The most common underlying and contributing causes of death in SCI patients are diseases of the circulatory and respiratory system.

It is recognised that weight gain is a common problem in patients with a SCI, typically occurring within the first year of rehabilitation and continuing life long. SCI patients have been shown to have an increased fat mass, waist circumference and altered lipid profile. Obesity in SCI patients can lead to an increased incidence of metabolic syndrome.

Patient weight gain is thought to be attributed to the reduction in energy expenditure compared to pre-injury levels, the loss of voluntary muscle use below the spinal cord lesion and reduction in lean tissue mass. It has been shown that the basal metabolic rate (BMR) of SCI patients is lower than predicted, with the greatest difference being for high tetraplegics. Findings suggest there is an overestimation of energy requirements in a small population of medically stable SCI patients. In addition, SCI calorie and protein intake is high in this patient population, suggesting that patients are also exceeding their nutritional recommendations. Excess calorie intake, reduction in energy requirement and / or a reduction in exercise will predispose the SCI patient to weight gain and obesity. Further understanding of this energy imbalance needs to be addressed.

This single centre feasibility study will initially determine if it is feasible to measure the 'actual' energy requirements of paraplegic and tetraplegic (ventilated and non-ventilated) in-patients during bed rest and rehabilitation following acute SCI. This preliminary data will be compared to 'predicted' energy expenditure levels. The calorie intake and body composition for each patient will be measured as well as factors indicative of metabolic syndrome. The study will initially provide statistical information in order to estimate the sample size required for a future definitive study on energy expenditure and development of metabolic syndrome in SCI patients. In addition, the feasibility study will address patient recruitment rates and reasons for withdrawal from the study and highlight any practicality issues with study conduct.

Recruitment:

15 acute paraplegic and 15 acute tetraplegic (ventilated and non-ventilated) inpatients will recruited.

Methodology:

The following procedures will be performed at bed rest, early mobilisation and hospital discharge:

Measurement of Actual Energy Expenditure Actual resting energy expenditure (REE) is determined by measuring the oxygen consumption and carbon dioxide production of a patient at rest using the GE Healthcare metabolic oxygenator. During the test, the individual is interfaced with a metabolic measurement system by means of a facemask. For ventilated patients, the monitor will be used with a cuffed tracheostomy tube.

Software will be used to calculate the respiratory quotient (RQ).

Calculating Predicted Energy Requirements Henry equations are used to predict the basal metabolic rate. Adjustments are made based on metabolic stress associated with illness and for obese individuals.

Determining Dietary Intake The patient's dietary intake will be reported using the standard hospital food charts. These will be completed for all food and fluids taken providing an indication of portion sizes. The charts will be kept for 3 consecutive days at each time point and is based on a pragmatic approach to improve accuracy of completion over a short period of time whilst still providing daily variations in intake. Data will be collected so that it covers at least one day of a weekend.

Anthropometric Measurements

Anthropometric measurements will be taken to determine patient body fat and muscle. The following parameters will be measured:

1. Mid Upper Arm Circumference (MUAC)
2. Tricep Skinfold Thickness (TSF)

Mid Arm Muscle Circumference (MAMC) will be calculated using the equation:

MAMC = MUAC - 3.14 x TSF

Metabolic Syndrome Measurements

The following will be measured:

1. Weight
2. Height
3. BMI Calculation
4. Blood Pressure
5. Waist Circumference
6. Fasting glucose, HDL, triglycerides

ELIGIBILITY:
Inclusion Criteria:

* Aged 18+ years old inclusive
* Traumatic and non-traumatic tetraplegic or paraplegic patient following acute SCI injury
* First referral to the Sheffield Spinal Injuries Centre
* Pressure ulcer(s) category 1 and/or 2 or normal skin
* Be able to provide written informed consent or verbal consent in the presence of an independent witness
* Ventilated patients without sedation
* Enterally fed patients

Exclusion Criteria:

* Aged less than 18 years old
* Lack the mental capacity to consent
* Pressure ulcer(s) category 3 and/or 4
* Previously had or currently have metabolic syndrome
* Previously had or currently have diabetes
* Current medication includes either a stimulant(s) and/or depressant(s) e.g. steroids, anti-depressants
* MRSA bacterium positive
* Previously had or currently has an eating disorder
* Ventilated patients with sedation
* Currently participating in another research study which may have an impact on the study or patient safety and well-being.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08-10 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Sample size for definitive study | 1 year
  Standard deviation of Resting Energy Expenditure measurements at hospital admission, initial mobilisation and hospital discharge

SECONDARY OUTCOMES:
Recruitment Period for Definitive Study | 1 year
  Number of patients recruited per year
Predicted Energy Requirements | 1 year
  Basal metabolic rate at hospital admission, initial mobilisation and hospital discharge
Dietary Intake | 1 year
  Hospital food chart analysis upon hospital admission, at initial mobilisation and hospital discharge
Muscle Measurements | 1 year
  Mid arm muscle circumference measured at hospital admission, initial mobilisation and hospital discharge
Adipose Tissue Measurements | 1 year
  Waist circumference measured at hospital admission, initial mobilisation and hospital discharge
Lipid Measurements | 1 year
  Fasting blood lipid profile measured at hospital admission, initial mobilisation and hospital discharge
BMI Measurements | 1 year
  BMI calculated from height and weight measurements at hospital admission, initial mobilisation and hospital discharge
Blood Pressure Measurements | 1 year
  Blood pressure measured at hospital admission, initial mobilisation and hospital discharge
Glucose Measurements | 1 year
  Fasting blood glucose measured at hospital admission, initial mobilisation and hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Northern General Hospital, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No